CLINICAL TRIAL: NCT06939491
Title: Comparison of Ultrasound-Guided Electrolysis Therapy (USGET) vs. Sham USGET on Patients With Patellar Tendinopathy: A Randomized Controlled Trial (RCT) Assessing the Effects on Pain, Function, and Tendon Structure Including MRI and Shear-wave Elastography Ultrasound Imaging
Brief Title: Comparison of Ultrasound-guided Electrolysis Therapy vs. Sham Electrolysis in Patients With Patellar Tendinopathy: A Prospective Randomized Study Including MRI and Shear-wave Ultrasound Elastography Imaging
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gymna Uniphy (Industry)
Collaborators: Paracelsus Klinik Bremen (Other); Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 898
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Patellar Tendinopathy / Jumpers Knee
Keywords: patellar tendinopathy; jumpers knee; ultra-sound-guided-electrolysis; electrolysis; galvanic current; USGET

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided galvanic electrolysis (USGET) (Experimental): The patients randomized in this group will receive the ultrasound-guided-electrolysis-therapy (acupuncture treatment including galvanic current, 5 applications at intervals of 2 weeks) + PTLE-Training protocol. Local peritendinous injection of the local anaesthetic mepivacaine (manufacturer: Puren, dosage: 10mg/ml, dose: 20mg (2ml), concentration: 1%) before performing electrolysis. The treatment period is 4 months, follow-up period totalling 3 months
  Interventions: Device: Ultrasound guided electrolysis therapy
- Sham Electrolysis (Sham Comparator): The patients randomized in this group will receive the sham-electrolysis with a current intensity of 0 mA (acupuncture treatment without galvanic current, 5 applications at intervals of 2 weeks) + PTLE-training protocol. Local peritendinous injection of the local anaesthetic mepivacaine (manufacturer: Puren, dosage: 10mg/ml, dose: 20mg (2ml), concentration: 1%) before performing sham electrolysis. The treatment period is 4 months, follow-up period totalling 3 months.
  Interventions: Device: Sham Electrolysis

INTERVENTIONS:
Device: Ultrasound guided electrolysis therapy — Ultrasound-guided galvanic electrolysis (USGET) is a technique most commonly used on chronically affected tissue. A galvanic current flows through an acupuncture needle producing an inflammatory reaction in the tissue. The inflammatory reaction will trigger a host of biological processes in the body. These will ultimately start the generation of new immature collagen fibres. The fibres become mature by means of training stimulus.
  The technique shows good results on tendons in the chronic phase, and may be used for injuries, such as long-standing muscle injury and treatment of myofascial pain syndrome and trigger points.
  Other Names: USGET
  Arms: Ultrasound-guided galvanic electrolysis (USGET)
Device: Sham Electrolysis — The same intervention as the electrolysis group with the device turned on but the current intensity turned to 0 mA (e.g., no galvanic current).
  Other Names: Sham Treatment
  Arms: Sham Electrolysis

SUMMARY:
Study Background and Purpose Tendinopathies are common and debilitating musculoskeletal disorders that often lead to chronic pain and reduced mobility. Traditional treatments face challenges due to limited tendon blood supply, leading to poor healing. This study investigates ultrasound-guided galvanic electrolysis therapy (USGET), which uses electric current to promote tendon healing, comparing its efficacy with a placebo.

Objectives The primary goal is to assess pain reduction, while secondary goals evaluate functionality, elasticity, and morphological changes (imaging) in patients with patellar tendinopathy.

Methodology

* Design: Prospective, randomized, double-blind, placebo-controlled study.
* Duration: 24 months (October 2024 - October 2026).
* Groups:
* Intervention Group: Electrolysis therapy with galvanic current, Progressive tendon-loading exercises.
* Control Group: Electrolysis placebo (without current), Progressive tendon-loading exercises.
* Sample Size: 74 subjects.
* Data Collection: Baseline, post-treatment (4 months), and follow-up (7 months).

Evaluation and Data Analysis The study assesses pain via VAS and functionality scores, alongside imaging (MRI, sonography) to measure tendon morphology. Statistical analysis includes hypothesis testing and regression using SPSS software.

Ethics and Publication Ethics approval is from the Bremen Medical Chamber. Results will be published regardless of outcome, following Good Clinical Practice and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 59 years,
* Informed consent (capable of giving consent),
* Presentation and diagnosis of patella tendinopathy without other concomitant musculoskeletal diseases or degenerative joint disease.

Exclusion Criteria:

* Children (< 18 years), age > 59 years,
* Pregnancy and breastfeeding,
* Patients who are unable to give consent,
* Musculoskeletal concomitant diseases such as fractures, sprains, dislocations, structural muscle injuries, meniscopathies, cruciate ligament injuries,
* Joint diseases (acute, degenerative) such as arthrosis or arthritis,
* Acute infections / open wounds in the area of the tendon to be examined
* Other relevant damage to the tendon to be examined
* Local steroid injections into the tendon before and after the start of the study,
* Injections of vascular sclerosing agents before and after the start of the study,
* Ingestion of fluoroquinolones, anticoagulants or anti-inflammatory drugs.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline to the end of treatment at 10 weeks
  The pain Visual Analogue Scale (VAS) is a subjective, unidimensional measure of pain intensity, used to record patients' pain progression. It is a horizontal line, 100 mm in length, that represent the severity of symptoms from 0 "no symptoms" to 10 "very severe symptoms." The patient marks on the line the point that the patient believes represents his or her perception of his or her current state.
Visual Analogue Scale (VAS) | Change from baseline to 7 months follow-up
  The pain Visual Analogue Scale (VAS) is a subjective, unidimensional measure of pain intensity, used to record patients' pain progression. It is a horizontal line, 100 mm in length, that represent the severity of symptoms from 0 "no symptoms" to 10 "very severe symptoms." The patient marks on the line the point that the patient believes represents his or her perception of his or her current state.

SECONDARY OUTCOMES:
Tegner Activity Scale | Change from baseline to the end of treatment at 10 weeks
  The Tegner Activity Scale (TAS) is a one-item score used to measure activity level, particularly in the context of knee injuries and sports. It uses a scale of 0 to 10, where 0 represents maximum disability and 10 represents participation in competitive sports at a national or international elite level.
Tegner Activity Scale | Change from baseline to 7 months follow-up
  The Tegner Activity Scale (TAS) is a one-item score used to measure activity level, particularly in the context of knee injuries and sports. It uses a scale of 0 to 10, where 0 represents maximum disability and 10 represents participation in competitive sports at a national or international elite level.
Visa-P | Change from baseline to the end of treatment at 10 weeks
  The Visa-P questionnaire (Victorian Institute of Sport Assessment - Patella) is a self-reported outcome measure that evaluates symptoms, function and the ability to play sports. The questionnaire consists of 8 questions designed to assess the patient's pain and functional ability during patellofemoral loading activities. The total score ranges from 0 to 100, with 100 representing an asymptomatic individual able to fully engage in sports and 0 representing the worst possible outcome.
Visa-P | Change from baseline to 7 months follow-up
  The Visa-P questionnaire (Victorian Institute of Sport Assessment - Patella) is a self-reported outcome measure that evaluates symptoms, function and the ability to play sports. The questionnaire consists of 8 questions designed to assess the patient's pain and functional ability during patellofemoral loading activities. The total score ranges from 0 to 100, with 100 representing an asymptomatic individual able to fully engage in sports and 0 representing the worst possible outcome.
International Knee Documentation Committee score | Change from baseline to the end of treatment at 10 weeks
  The International Knee Documentation Committee score (IKDC) is a tool used to assess knee function and symptoms. It's a patient-completed questionnaire that helps quantify how a person's knee is affecting their daily activities and sports participation. The score ranges from 0 to 100, with higher scores indicating better function and fewer symptoms.
International Knee Documentation Committee score | Change from baseline to 7 months follow-up
  The International Knee Documentation Committee score (IKDC) is a tool used to assess knee function and symptoms. It's a patient-completed questionnaire that helps quantify how a person's knee is affecting their daily activities and sports participation. The score ranges from 0 to 100, with higher scores indicating better function and fewer symptoms.
Comprehensive Aachen Knee Score | Change from baseline to the end of treatment at 10 weeks
  The Comprehensive Aachen Knee Score (COMPACK) is a novel, reliable and valid instrument to measure knee pain regarding two dimensions, intensity and frequency from the patient perspective. The total score consist of two subscales and ranges from 0 (no pain or frequency of pain) to 60 (the worst possible pain and pain frequency).
Comprehensive Aachen Knee Score | Change from baseline to 7 months follow-up
  The Comprehensive Aachen Knee Score (COMPACK) is a novel, reliable and valid instrument to measure knee pain regarding two dimensions, intensity and frequency from the patient perspective. The total score consist of two subscales and ranges from 0 (no pain or frequency of pain) to 60 (the worst possible pain and pain frequency).
B-scan sonography | Change from baseline to the end of treatment at 10 weeks
  B-scan sonography, or ultrasound imaging, is a valuable tool for assessing tendon conditions. It allows visualization of tendon structure, dimensions, and potential pathologies like tears or inflammation. B-mode ultrasound can show the fibrillar pattern of normal tendons and help identify abnormalities, such as the presence of tears or the degree of tendon retraction in cases of rupture
B-scan sonography | Change from baseline to 7 months follow-up
  B-scan sonography, or ultrasound imaging, is a valuable tool for assessing tendon conditions. It allows visualization of tendon structure, dimensions, and potential pathologies like tears or inflammation. B-mode ultrasound can show the fibrillar pattern of normal tendons and help identify abnormalities, such as the presence of tears or the degree of tendon retraction in cases of rupture
Doppler sonography | Change from baseline to the end of treatment at 10 weeks
  Doppler sonography, a type of ultrasound, is used to assess blood flow within tendons, particularly in conditions like tendinopathy or tendinosis. It can help visualize neovascularization (new blood vessel formation) within abnormal tendons.
Doppler sonography | Change from baseline to 7 months follow-up
  Doppler sonography, a type of ultrasound, is used to assess blood flow within tendons, particularly in conditions like tendinopathy or tendinosis. It can help visualize neovascularization (new blood vessel formation) within abnormal tendons.
Shear wave elastography | Change from baseline to the end of treatment at 10 weeks
  Shear wave elastography (SWE) is a non-invasive ultrasound technique that can be used to assess tendon stiffness and elasticity. It measures the speed of shear waves as they travel through the tendon, which can be related to the tissue's mechanical properties. SWE can help differentiate between healthy and pathological tendons, potentially aiding in the diagnosis and monitoring of tendinopathies
Shear wave elastography | Change from baseline to 7 months follow-up
  Shear wave elastography (SWE) is a non-invasive ultrasound technique that can be used to assess tendon stiffness and elasticity. It measures the speed of shear waves as they travel through the tendon, which can be related to the tissue's mechanical properties. SWE can help differentiate between healthy and pathological tendons, potentially aiding in the diagnosis and monitoring of tendinopathies
Magnetic resonance imaging | Change from baseline to the end of treatment at 10 weeks
  Magnetic resonance imaging (MRI) can be used to assess tendinopathy, by detecting structural changes and inflammatory processes. It's particularly useful for evaluating partial tears and postoperative assessment, offering better visualization than ultrasound in these situations. MRI can also identify other associated injuries like cartilage damage, bone abnormalities, and ligament injuries
Magnetic resonance imaging | Change from baseline to 7 months follow-up
  Magnetic resonance imaging (MRI) can be used to assess tendinopathy, by detecting structural changes and inflammatory processes. It's particularly useful for evaluating partial tears and postoperative assessment, offering better visualization than ultrasound in these situations. MRI can also identify other associated injuries like cartilage damage, bone abnormalities, and ligament injuries

CONTACTS AND LOCATIONS:
Locations (1):
- Paracelsus Sportmedizin & Prävention Bremen, Bremen, City state Bremen, Germany

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: 01.08.2026 until 31.12.2026

REFERENCES:
- [Background] Risch L, Wochatz M, Messerschmidt J, Engel T, Mayer F, Cassel M. Reliability of Evaluating Achilles Tendon Vascularization Assessed With Doppler Ultrasound Advanced Dynamic Flow. J Ultrasound Med. 2018 Mar;37(3):737-744. doi: 10.1002/jum.14414. Epub 2017 Sep 28. PMID 28960372
- [Background] Krott NL, Wild M, Betsch M. The Comprehensive Aachen Knee Score: Development and validation of a new patient-reported outcome measure for patellofemoral pathologies. Knee. 2021 Oct;32:112-120. doi: 10.1016/j.knee.2021.08.010. Epub 2021 Aug 27. PMID 34461387
- [Background] Higgins LD, Taylor MK, Park D, Ghodadra N, Marchant M, Pietrobon R, Cook C; International Knee Documentation Committee. Reliability and validity of the International Knee Documentation Committee (IKDC) Subjective Knee Form. Joint Bone Spine. 2007 Dec;74(6):594-9. doi: 10.1016/j.jbspin.2007.01.036. Epub 2007 Aug 6. PMID 17888709
- [Background] Hernandez-Sanchez S, Hidalgo MD, Gomez A. Responsiveness of the VISA-P scale for patellar tendinopathy in athletes. Br J Sports Med. 2014 Mar;48(6):453-7. doi: 10.1136/bjsports-2012-091163. Epub 2012 Sep 25. PMID 23012320
- [Background] Tegner Y, Lysholm J. Rating systems in the evaluation of knee ligament injuries. Clin Orthop Relat Res. 1985 Sep;(198):43-9. PMID 4028566
- [Background] Larrivee S, Balg F, Leonard G, Bedard S, Tousignant M, Boissy P. Wrist-Based Accelerometers and Visual Analog Scales as Outcome Measures for Shoulder Activity During Daily Living in Patients With Rotator Cuff Tendinopathy: Instrument Validation Study. JMIR Rehabil Assist Technol. 2019 Dec 3;6(2):e14468. doi: 10.2196/14468. PMID 31793896
- [Background] Ito N, Sigurethsson HB, Pohlig RT, Cortes DH, Gravare Silbernagel K, Sprague AL. Reliability of Continuous Shear Wave Elastography in the Pathological Patellar Tendon. J Ultrasound Med. 2023 May;42(5):1047-1055. doi: 10.1002/jum.16115. Epub 2022 Oct 27. PMID 36301665
- [Background] Abat F, Alfredson H, Cucchiarini M, Madry H, Marmotti A, Mouton C, Oliveira JM, Pereira H, Peretti GM, Spang C, Stephen J, van Bergen CJA, de Girolamo L. Current trends in tendinopathy: consensus of the ESSKA basic science committee. Part II: treatment options. J Exp Orthop. 2018 Sep 24;5(1):38. doi: 10.1186/s40634-018-0145-5. PMID 30251203
- [Background] Asensio-Olea L, Leiros-Rodriguez R, Marques-Sanchez MP, de Carvalho FO, Maciel LYS. Efficacy of percutaneous electrolysis for the treatment of tendinopathies: A systematic review and meta-analysis. Clin Rehabil. 2023 Jun;37(6):747-759. doi: 10.1177/02692155221144272. Epub 2022 Dec 30. PMID 36583575
- [Background] Dufner A, Thomas G. Ribosomal S6 kinase signaling and the control of translation. Exp Cell Res. 1999 Nov 25;253(1):100-9. doi: 10.1006/excr.1999.4683. PMID 10579915
- [Background] Eliasson J, Elfegoun T, Nilsson J, Kohnke R, Ekblom B, Blomstrand E. Maximal lengthening contractions increase p70 S6 kinase phosphorylation in human skeletal muscle in the absence of nutritional supply. Am J Physiol Endocrinol Metab. 2006 Dec;291(6):E1197-205. doi: 10.1152/ajpendo.00141.2006. Epub 2006 Jul 11. PMID 16835402
- [Background] Lepley LK, Stoneback L, Macpherson PCD, Butterfield TA. Eccentric Exercise as a Potent Prescription for Muscle Weakness After Joint Injury. Exerc Sport Sci Rev. 2023 Jul 1;51(3):109-116. doi: 10.1249/JES.0000000000000319. Epub 2023 Apr 24. PMID 37093645
- [Background] Penin-Franch A, Garcia-Vidal JA, Martinez CM, Escolar-Reina P, Martinez-Ojeda RM, Gomez AI, Bueno JM, Minaya-Munoz F, Valera-Garrido F, Medina-Mirapeix F, Pelegrin P. Galvanic current activates the NLRP3 inflammasome to promote Type I collagen production in tendon. Elife. 2022 Feb 24;11:e73675. doi: 10.7554/eLife.73675. PMID 35199642
- [Background] Muaidi QI. Rehabilitation of patellar tendinopathy. J Musculoskelet Neuronal Interact. 2020 Dec 1;20(4):535-540. PMID 33265081
- [Background] Riel H, Lindstrom CF, Rathleff MS, Jensen MB, Olesen JL. Prevalence and incidence rate of lower-extremity tendinopathies in a Danish general practice: a registry-based study. BMC Musculoskelet Disord. 2019 May 22;20(1):239. doi: 10.1186/s12891-019-2629-6. PMID 31113484
- [Background] Lian OB, Engebretsen L, Bahr R. Prevalence of jumper's knee among elite athletes from different sports: a cross-sectional study. Am J Sports Med. 2005 Apr;33(4):561-7. doi: 10.1177/0363546504270454. Epub 2005 Feb 8. PMID 15722279
- [Background] Kujala UM, Sarna S, Kaprio J. Cumulative incidence of achilles tendon rupture and tendinopathy in male former elite athletes. Clin J Sport Med. 2005 May;15(3):133-5. doi: 10.1097/01.jsm.0000165347.55638.23. PMID 15867554
- [Background] Hopkins C, Fu SC, Chua E, Hu X, Rolf C, Mattila VM, Qin L, Yung PS, Chan KM. Critical review on the socio-economic impact of tendinopathy. Asia Pac J Sports Med Arthrosc Rehabil Technol. 2016 Apr 22;4:9-20. doi: 10.1016/j.asmart.2016.01.002. eCollection 2016 Apr. PMID 29264258
- [Background] Graca AL, Gomez-Florit M, Gomes ME, Docheva D. Tendon Aging. Subcell Biochem. 2023;103:121-147. doi: 10.1007/978-3-031-26576-1_7. PMID 37120467
- [Background] Mirghaderi SP, Valizadeh Z, Shadman K, Lafosse T, Oryadi-Zanjani L, Yekaninejad MS, Nabian MH. Cell therapy efficacy and safety in treating tendon disorders: a systemic review of clinical studies. J Exp Orthop. 2022 Aug 30;9(1):85. doi: 10.1186/s40634-022-00520-9. PMID 36042110
- [Background] Abat F, Sanchez-Sanchez JL, Martin-Nogueras AM, Calvo-Arenillas JI, Yajeya J, Mendez-Sanchez R, Monllau JC, Gelber PE. Randomized controlled trial comparing the effectiveness of the ultrasound-guided galvanic electrolysis technique (USGET) versus conventional electro-physiotherapeutic treatment on patellar tendinopathy. J Exp Orthop. 2016 Dec;3(1):34. doi: 10.1186/s40634-016-0070-4. Epub 2016 Nov 16. PMID 27854082
- See also: The Acure 8000 is the device used for the ultrasound-guided-electrolysis therapy — https://gymna.com/de/produkte/electrolysis/gymna-acure-8000/gymna-acure-8000